CLINICAL TRIAL: NCT00002446
Title: Randomized, Controlled Trial of SCH 56592 Oral Suspension Versus Fluconazole Suspension in the Treatment of Oropharyngeal Candidiasis (OPC) in HIV-Positive Patients
Brief Title: Safety and Effectiveness of Fluconazole Versus SCH 56592 to Treat Thrush in HIV-Positive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Schering-Plough (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 305A; C97-331; I97-331
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-02

CONDITIONS: Candidiasis, Oral; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Fluconazole; Administration, Oral; Antifungal Agents; Candidiasis, Oral; Pharyngeal Diseases; posaconazole
MeSH Terms: conditions — Candidiasis, Oral; HIV Infections; AIDS-Related Opportunistic Infections; Pharyngeal Diseases | interventions — posaconazole; Fluconazole

INTERVENTIONS:
Drug: Posaconazole
Drug: Fluconazole

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of 2 treatments for thrush (a fungal infection of the mouth and throat) in HIV-positive patients. Fluconazole is a drug that is commonly used to treat thrush. SCH 56592 is a new drug that will be compared to fluconazole.

DETAILED DESCRIPTION:
Patients receive SCH 56592 oral suspension or fluconazole suspension for 14 days. Patients remain on study for 44 days total and are monitored for safety and efficacy of study treatment.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are at least 18 years old.
* Are HIV-positive.
* Have thrush (oropharyngeal candidiasis).
* Agree to practice sexual abstinence or use effective barrier methods of birth control (e.g., condoms).
* Are able to take study medication and return for clinic visits during the study.
* Are expected to live for at least 2 months.

Exclusion Criteria

You will not be eligible for this study if you:

* Have received protease inhibitors for the first time within 30 days prior to study entry.
* Have received certain medications.
* Have certain other types of fungal infections.
* Have certain types of cancer.
* Have received SCH 56592 within 3 months prior to study entry.
* Are pregnant or breast-feeding.
* Cannot take medications by mouth.
* Are allergic to azole drugs.
* Have certain medical conditions.
* Have been in this study before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1998-08

CONTACTS AND LOCATIONS:
Locations (18):
- United States (17):
  - East Bay AIDS Ctr, Berkeley, California
  - ViRx Inc, San Francisco, California
  - Kaiser Foundation Hospital, San Francisco, California
  - Infectious Disease and AIDS Clinic, Denver, Colorado
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Boulevard Comprehensive Care Ctr, Jacksonville, Florida
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - TRIAD Health Practice, Chicago, Illinois
  - Community Hosp Indianapolis, Indianapolis, Indiana
  - Wayne State Univ / Harper Hosp, Detroit, Michigan
  - UMDNJ - New Jersey Med School / Cooper Hosp, Camden, New Jersey
  - Jersey City Med Ctr, Jersey City, New Jersey
  - SUNY / Health Science Ctr at Brooklyn, Brooklyn, New York
  - Univ of Pennsylvania School of Dental Medicine, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Amelia Ct Clinic, Dallas, Texas
  - Univ of Texas Health Sciences Ctr, San Antonio, Texas
- Queen Elizabeth Hosp Respiratory Unit, Saint Michael, Barbados